CLINICAL TRIAL: NCT02013102
Title: A Randomized, Controlled, Multi-center Collaborative Phase Ⅳ Study to Evaluate the Safety and Efficacy of Decitabine in Myelodysplastic Syndrome
Brief Title: A Phase Ⅳ Study of Decitabine in Myelodysplastic Syndrome
Acronym: DREAM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cttq (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DREAM-201
Record Dates: First submitted 2013-12-09; First posted 2013-12-17 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm Ⅰ (Experimental): Decitabine Injection 20mg/m2/d*5d, IV> 1h, one cycles per 4 weeks.
  Interventions: Drug: Decitabine Injection
- Arm Ⅱ (Experimental): Decitabine Injection 12mg/m2/d*8d, IV> 1h, one cycles per 4 weeks.
  Interventions: Drug: Decitabine Injection

INTERVENTIONS:
Drug: Decitabine Injection — Decitabine Injection 20mg/m2/d*5d, IV> 1h, one cycles per 4 weeks; Decitabine Injection 12mg/m2/d*8d, IV> 1h, one cycles per 4 weeks.
  Other Names: qingweike

SUMMARY:
The purpose of this study is to evaluate of the safety and efficacy of decitabine treatment of Myelodysplastic Syndrome.

DETAILED DESCRIPTION:
Total subjects: 240, doseⅠgroup of 120 patients, doseⅡgroup of 120 patients. Subjects are stratified randomize. If necessary, participants accepted best supportive therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18;
* The diagnosis of MDS patients comply WHO2008 standards;
* IPSS score≥0.5;
* WHO classification for patients RCUD, RARS and transfusion-dependent RCMD;
* ECOG PS score: 0-2;
* Expected survival≥3 months;
* Serum bilirubin≤1.5*ULN, serum ALT and AST≤2.5*ULN, serum Cr≤1.5*ULN;
* Subjects signed informed consent form in line with GCP requirements.

Exclusion Criteria:

* Can not marrow biopsy;
* Previously diagnosed AML;
* Received azacitidine or decitabine treatment any time before;
* Being diagnosed with other malignancies in the prior 12 months;
* Pregnant or lactating women;
* Failure to control systemic fungal, bacterial or viral infection;
* Known or suspected allergy to decitabine;
* Known human immunodeficiency virus (HIV) or hepatitis B or C classes of active viral infection;
* Have a history of neurological or psychiatric disorders, including epilepsy or dementia;
* CTCAE 3 or 4 degree peripheral neuropathy;
* According to the investigator's judgment, there are concomitant diseases with a serious safety hazard or affect the patients completed the study in patients;
* Using other experimental drugs or participating in other clinical trials in the prior one months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The safety and efficacy of decitabine treatment of Myelodysplastic Syndrome. | 2-4 months
  The primary efficacy evaluation: ORR The secondary efficacy evaluation: CR，mCR，PR，HI, PFS in one year, Cytogenetic response, transfusion requirements, et al.

CONTACTS AND LOCATIONS:
Overall Officials: Shao Zonghong, MD, Principal Investigator — Tianjin Medical University General Hospital
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China